CLINICAL TRIAL: NCT05183165
Title: Description of the Copper Concentration in Breast Milk in Women Treated for Wilson's Disease
Acronym: WILLACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AOA_2021_28
Record Dates: First submitted 2021-12-21; First posted 2022-01-10 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Wilson's Disease
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Wilson's disease declaring pregnancy, (Other): Patients with Wilson's disease declaring pregnancy.Followed in the reference, constituent, and competence centers for Wilson's disease and other rare copper-related diseases, spread over French national territory.
  Interventions: Other: Patients with Wilson's disease declaring pregnancy,

INTERVENTIONS:
Other: Patients with Wilson's disease declaring pregnancy, — Blood and urine biological assessment Dietary assessment

SUMMARY:
Wilson's disease is a rare genetic disease, affecting less than 1,500 people in France. The transmission is autosomal recessive linked to an anomaly of the ATP7B gene on chromosome.This gene codes for an ATPase-type transmembrane protein involved in the transport of copper through the cell plasma member.This gene codes for an ATPase-type transmembrane protein involved in the transport of copper through the cell plasma member. If there is no mutation, this ATPase incorporates copper into apo-ceruloplasmin to be released into the blood serum. The mutation of the ATP7B gene results in a defective biliary excretion of copper, leading to its accumulation in the liver, but also in other organs such as the eye or the brain. Advances in treatment have dramatically changed the prognosis for Wilson's disease, making the desire for pregnancy more confident.

The consensus is to maintain treatment during pregnancy, reducing the dosage to limit teratogenicity as well as the risk of fetal copper deficiency.The mammary gland is the primary site of copper metabolism in lactation, and ATPase 7B is the primary effector.

It has been shown in a mouse model of Wilson's disease (ATP7B - / - mouse) with treatment, that mothers accumulate copper in the liver but also in the mammary gland.

However, a recent study showed that the copper level in breast milk was normal in 18 Wilsonian patients treated with D-penicillamine, trientine salts or zinc salts, suggesting that breastfeeding is possible in these patients without risk to the development of the infants.The problem of breastfeeding newborns for patients with Wilson's disease is therefore associated with a risk of copper deficiency in the newborn due to insufficiently rich breast milk in copper due to drugs.

In addition, the passage into breast milk of treatments is not sufficiently known.

These factors make breastfeeding not currently recommended for Wilsonian mothers,However, many patients wish to breastfeed and some of them breastfeed their newborns despite the risk of breastfeeding

ELIGIBILITY:
Criteria for inclusion :

* Patient aged 18 years or over.
* Wilson's disease fulfilling the criteria for the Leipzig score
* Pregnancy in progress whatever the term.
* Express consent to participate in the study.
* Affiliate or beneficiary of a social security system.

Criteria for non-inclusion :

* Liver transplant patient
* No affiliation to Social Security system
* VuInability to give free and informed consent
* Patient benefiting from a legal protection measure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-11 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Concentration of total copper (bound and free) in µmol / L in a sample of breast milk | 1 day ± 24 hours after childbirth
  The assay is performed by induced plasma mass spectrometry (ICP-MS) after nitric acid mineralization of the sample.
  Concentration of total copper (bound and free) in µmol / L in a sample of breast milk taken 1 day ± 24 hours after childbirth.
  The copper assay is performed by induced plasma mass spectrometry (ICP-MS) after nitric acid mineralization of the sample.
  The copper assay is performed by induced plasma mass spectrometry (ICP-MS) after nitric acid mineralization of the sample.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Adolphe de Rothschild, Paris, France